CLINICAL TRIAL: NCT03299881
Title: Safety and Effectiveness of Transcutaneous Electrical Nerve Stimulation (TENS)-Assisted Weight Loss
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to technical problems with the device.
Sponsor: Elira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-004
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, adaptive parallel arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): The Transcutaneous Nerve Stimulator (TENS) Elira wearable patch system will be applied to varying locations on the T6/T7 dermatone for 30 minutes three times a day after meals. Subjects will be instructed to follow a 1200 calorie healthy diet and record any changes in appetite.
  Interventions: Device: Transcutaneous Nerve Stimulator (TENS); Behavioral: Diet & Exercise
- Control (Active Comparator): Open label diet and exercise counseling only. Subjects will be instructed to follow a healthy 1200 calorie diet and record any changes in appetite.
  Interventions: Behavioral: Diet & Exercise

INTERVENTIONS:
Device: Transcutaneous Nerve Stimulator (TENS) — The Elira wearable patch system is a RF coupled, wearable transcutaneous electrical nerve stimulator (TENS) device controlled via Bluetooth by a smart phone unit running a custom application which directs therapy from the patch within safe limits set by a clinician and also includes a weight loss diary.
  Arms: Treatment
Behavioral: Diet & Exercise — Subjects to be instructed on a healthy 1200 calorie diet.

SUMMARY:
This study is a randomized, adaptive, parallel arm study. The treatment group will receive the Elira wearable patch system and provided instructions for use and advised to follow a 1200 calorie diet. The control group will be asked to follow a 12 calorie diet only. Each group will be followed for 12 weeks. Total body weight loss will be measured as well as appetite changes. Safety data will be collected throughout the study period. Safety and effectiveness will be determined based on differences between the groups.

DETAILED DESCRIPTION:
This study employs a randomized, adaptive, parallel arm study in which, cohorts of enrolled subjects (25 per arm) are assessed for dose response and progression to achievement of primary and secondary endpoints. Enrollment will be up to 300 subjects at 4 US centers.

After signing informed consent, subjects will be screened during a one week screening/baseline period to determine if they meet the inclusion criteria and exhibit none of the exclusion criteria. Weight, blood pressure, blood lipids, HgA1c, pregnancy test (for women of childbearing age), and patient questionnaires will be collected. If eligible, subjects will be randomized to treatment or control groups. The treatment group will receive training on the Elira Wearable Patch System and the first TENS session will be administered in the investigators office. Both groups will receive an electronic scale and instructions on 1200 calorie diet as well as diary completion requirements to be completed throughout the study. All subjects will be required to have in office follow-up visits every 4 weeks for 12 weeks. Up to 2 additional follow-up visits will be permitted within that 12 week time period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 - 65 years of age inclusive.
2. Subject has a BMI of 25-35 kg/ m^2 inclusive.
3. Subject has signed the informed consent form and is able to comply with study protocol and adhere to study visit schedule.
4. Subject is able to wear and use a wearable, patch TENS system.
5. Subject is able to use a touch screen hand held smart phone.
6. Subject is fluent in English and can complete patient questionnaires.
7. Subject can comply with a 1200 calorie the recommended diet for the duration of the study.
8. Subject is male or non-pregnant, non-lactating female, who agrees to use effective contraceptive methods throughout the length of the trial based on PI approval.
9. Females of childbearing potential must have a negative urine pregnancy test at enrollment visit, prior to placement of ELIRA device.

Exclusion Criteria

1. Subject has any known gastrointestinal disorder that in the opinion of the PI precludes enrollment into the trial.
2. Subject has had a prior bariatric procedure.
3. Subject has any significant multisystem disease in the opinion of the PI.
4. Subject has > 6.5 HbA1c.
5. Subject has significant cardiac arrhythmia, ectopy, or significant cardiovascular disease.
6. Subject has an existing implanted electrical stimulator (e.g., pacemaker, AICD).
7. Subject is a female of child-bearing potential who is pregnant or intends to become pregnant during the trial.
8. Subject has a history of any malignancy in the last 2 years.
9. Subject has had a weight change of + 5% of his/her Total Body Weight in the 3 months prior to enrollment.
10. Subject has a moderate / severe psychiatric disorder.
11. Subject has a diagnosed neurological disease.
12. Subject has a diagnosed eating disorder.
13. Subject has a skin disorder affecting the thoracic dermatomes.
14. Subject has abdominal surgery or other scars which may interfere with stimulation in the opinion of the PI.
15. Subject is currently enrolled in other, potentially confounding research.
16. Subject has known allergic reaction to materials in the electrodes and/or is otherwise unable to tolerate stimulation with the wearable TENS system.
17. Subject is actively participating or unwilling to discontinue participation in another weight loss program.
18. Subject is taking weight loss control medications including but not limited to OTC medications, Metformin, and Belviq.
19. Subject is unable to take anti-nausea medications planned for the study.
20. Inability to walk at least 0.8 kilometers per day (10 minutes of continuous walking).
21. Current smoker or user of nicotine product or smoking cessation within 1 year of the screening date.
22. History of treatment for or current abuse of drugs or alcohol.
23. A score of ≥10 on the Patient Health Questionnaire 9 (PHQ-9), demonstrating moderate depression.
24. Any subject that the investigator considers inappropriate for the study for medical reasons.
25. Subject has a history of migraine and/or is taking Topiramate for severe headache disorders.
26. Subject is on hormonal or other drug therapy which may alter antral motility or appetite, per physician discretion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Sullivan, MD, Principal Investigator — Consultant
Locations (1):
- St. Louis Women's Healthcare Group, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 39 | 38
Completed | 22 | 25
Not Completed | 17 | 13
Not completed — Study Termination | 17 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Full Range); unit: years] | 48.2 [28 to 65] | 46.5 [19 to 64] | 47.4 [19 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 2 | 3 | 5
  Race/Ethnicity: White | 36 | 35 | 71
  Race/Ethnicity: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77
BMI [Mean (Full Range); unit: kg/m^2] | 29.9 [26.3 to 34.5] | 29.2 [25.4 to 34.5] | 29.6 [25.4 to 34.5]
Weight [Mean (Full Range); unit: pounds] | 178.5 [142.6 to 220.2] | 174.6 [149.4 to 200.2] | 176.6 [142.6 to 220.2]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: Safety/Tolerability will be assessed by the non-inferiority of incidence of serious adverse events (SAEs), unanticipated DAEs (USAEs), device-related SAEs (DSAEs), and unanticipated device-related SAEs (UDAEs) that are associated with the TENS therapy throughout the stimulation and the follow-up period versus historical control (compared with other TENS systems).
Time Frame: 12 weeks
Population: Study was terminated and recruitment was stopped. Sincere efforts were made but technical difficulties with device prevented the necessary data collection to allow specified outcome analysis. Adverse event data is reported.
Measure: Number; unit: Serious Adverse Events
Arm/Group | Treatment | Control
Number analyzed (Participants) | 39 | 38
Serious Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 39/39 | 23/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=39) | Control (N=38)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Blistering rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Worsening contact dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Body rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 6 (6) | 2 (2)
Intraductal papilloma mass, left breast (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1)
Poison ivy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cracked tooth (General disorders) | 1 (1) | 0 (0)
Torn rotator cuff (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Strep throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Swelling, upper extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bartholin's gland abscess (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Left knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Venous thoracic outlet syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to technical problems with the device. Insufficient data to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT03299881/Prot_SAP_000.pdf